CLINICAL TRIAL: NCT05704348
Title: A Clinical Intervention Study Exploring Gastropexy as a Measure to Reduce Gastro-oesophageal Reflux Disease After Laparoscopic Sleeve Gastrectomy
Brief Title: Sleeve-pex: A Randomized Trial to Reduce Reflux After Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Forde (Other)
Responsible Party: Principal Investigator, Villy Våge, Project leader, Helse Forde
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 421917
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Gastropexy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The patient and the healtcare workers will be masked as to whether a pexi has been performed or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No gastropexy (Active Comparator): Sleeve gastrectomy without gastropexy.
  Interventions: Procedure: Sleeve gastrectomy without gastropexy
- Gastropexy (Experimental): Sleeve gastrectomy with gastropexy
  Interventions: Procedure: Sleeve gastrectomy with gastropexy

INTERVENTIONS:
Procedure: Sleeve gastrectomy with gastropexy — Gastropexy in this project means suturing the gastric remnant to the gastrocolic ligament.
  Arms: Gastropexy
Procedure: Sleeve gastrectomy without gastropexy — Sleeve gastrectomy without suturing the gastric remnant to the gastrocolic ligament.
  Arms: No gastropexy

SUMMARY:
The goal of this clinical trial is to test gastropexy as a measure to reduce reflux in morbidly obese patients being submitted to sleeve gastrectomy. The main questions it aims to answer are:

Does gastropexy reduce reflux symptoms? Does gastropexy reduce objective evidence of reflux? Participants will be randomized to gastropexy or no gastropexy, and researchers will compare these groups to see if reflux (symptoms / objective evidence of) is different in the two groups.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy (LSG) has become the most commonly performed bariatric procedure worldwide. LSG consists of a longitudinal resection of the stomach leaving the intestines intact, thereby lowering the risk for side-effects due to rerouting of the small bowel. However, gastro-esopageal reflux disease (GERD) has been reported to increase after LSG. Our hypothesis is that GERD is mainly due to intrathoracic migration of the gastric remnant. The aim of this study is to explore if suturing the gastric remnant to the gastrocolic ligament (gastropexy) will prevent intrathoracic migration and thereby reduce the development of reflux.

Patients planned for a sleeve gastrectomy will be invited to participate, and participating patients will be randomized to pexi or no pexi. According to power calculations a total of 550 patients will be randomized in the study. Follow-up will be at six weeks, one-, two- and five years.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for bariatric surgery with primary LSG

Exclusion Criteria:

* Age below 18 yrs
* Use of ARM for other reasons than reflux
* Previous antireflux surgery
* Inability to comprehend and respon to patient related outcome (PRO) questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2023-09-04 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants using acid-reducing medication (ARM) or having had reoperations due to GERD | Two years
  ARM: Daily use of ARM for the last month

SECONDARY OUTCOMES:
Endoscopic findings | Two years
  Visible oesophagitis according to the LA classification
Patient related outcome | Two years
  GerdQ questionnaire
pH-metry | Two years
  pH measurement by Bravo capsule

CONTACTS AND LOCATIONS:
Overall Officials: Villy Vage, MD PhD, Study Chair — Helse Forde
Locations (4):
- Norway (4):
  - Helse Forde, Førde
  - Aleris Oslo, Oslo
  - Volda sjukehus, Volda
  - Voss sjukehus, Voss

IPD SHARING:
Plan to Share IPD: Yes
Information about Sleeve-pex will be found at the SOReg-N webpage.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol including analysis plan and formula for informed consent will be available at the SOReg-N webpage from the beginning of the study.
Access Criteria: The study protocol is available at SOReg-N webpage. Data from the study will be made available for other researchers on request if approved by the ethical review board.
URL: https://helse-bergen.no/avdelinger/laboratorieklinikken/medisinsk-biokjemi-og-farmakologi/norsk-kvalitetsregister-for-fedmekirurgi-soreg-norge